CLINICAL TRIAL: NCT04294914
Title: Catastrophizing and Virtual Reality's Impact on the Pain Threshold During a Cold Pressor Test in Patients With Fibromyalgia: A Case-control Study
Brief Title: Catastrophizing and Virtual Reality's Impact on Pain in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Naestved Hospital (Other)
Responsible Party: Principal Investigator, Steffan Wittrup Christensen, Associate professor, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SJ-822
Record Dates: First submitted 2020-02-29; First posted 2020-03-04 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Fibromyalgia; Pain
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Intervention Model Description: Half the participants will start with intervention 1 after which they will crossover to intervention 2. The other half will start start with intervention 2 before crossing over to intervention 1.
Who Masked: Participant
Masking Description: The participants are blind to the study hypothesis and therefore the expected outcome of the tests performed
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibromyalgia (Active Comparator): Individuals with fibromyalgia.
  Interventions: Other: Cold Pressor Test; Other: Cold Pressor Test + Virtual Reality
- Healthy controls (Experimental): Healthy, pain-free individuals
  Interventions: Other: Cold Pressor Test; Other: Cold Pressor Test + Virtual Reality

INTERVENTIONS:
Other: Cold Pressor Test — The participant submerges one limb into a tank of cold (1-2 ° C), circulating water.
Other: Cold Pressor Test + Virtual Reality — The participant submerges one limb into a tank of cold (1-2 ° C), circulating water while interacting with a virtual reality environment

SUMMARY:
This study evaluates the potential association between Virtual Reality, pain catastrophizing thoughts and pain measures in fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand, read and speak Danish
* Able to independently answer a questionnaire
* Able to give informed consent

Fibromyalgia group:

* Confirmed diagnosed with fibromyalgia

Controls:

* Healthy participants

Exclusion Criteria:

Applies for both groups:

* Signs of anxiety, depression and post-traumatic stress syndrome that require treatment
* Neurologic, musculoskeletal or mental illnesses that could influence the results.
* Parallel participating in other studies, that can influence this study
* Pregnancy

Fibromyalgia group:

* Regulation in medication
* Anticonvulsivant use the last week
* Serotonin-norepinephrine reuptake Inhibitor (SNRI) the last two weeks
* Tricykliske antidepressants (TCA) the last four weeks

Controls:

* No regular use of pain medication
* No current or previous history of subacute or ongoing pain

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity | through study completion, an average of 90minutes
  Pain intensity during the interventions is scored using a Visual Analog Scale or Numeric Rating Scale (0 = no pain and 10 = worst known pain)
Pain threshold | through study completion, an average of 90minutes
  Pain threshold is defined as when the participants feel the sensation changing from an unpleasant feeling to a painful experience (measured in seconds)
Pain tolerance | through study completion, an average of 90minutes
  Pain tolerance is when the participants no longer are able to withstand the pain (measured in seconds).

SECONDARY OUTCOMES:
Pain catastrophizing | through study completion, an average of 90minutes
  The pain catastrophizing score is measured by filling out the pain catastrophizing scale questionnaire. The pain catastrophizing scale consists of 13 sentences assessing pain-related thoughts or feelings. These are then divided into 3 domains: rumination, magnification and helplessness. The subject is asked to rate how well each sentence applies for them: 0 = not at all, 1 = to a slight degree, 2 = to a moderate degree, 3 = to a great degree and 4 = all the time.
  The total score on the questionnaire can lie between 0 - 52 where a higher score indicates higher levels of pain catastrophizing thoughts.

CONTACTS AND LOCATIONS:
Overall Officials: Steffan WM Christensen, PhD, Principal Investigator — Dept. Of Health Science and Technology, Aalborg University
Locations (1):
- Interdisciplinary Paincenter Naestved, Naestved hospital, Næstved, Region Sjælland, Denmark

REFERENCES:
- [Derived] Christensen SWM, Almsborg H , M, Vain TS , M, Vaegter HB. The Effect of Virtual Reality on Cold Pain Sensitivity in Patients with Fibromyalgia and Pain-Free Individuals: A Randomized Crossover Study. Games Health J. 2023 Aug;12(4):295-301. doi: 10.1089/g4h.2022.0138. Epub 2022 Nov 28. PMID 36454199